CLINICAL TRIAL: NCT06664684
Title: Effects of Intermittent Fasting in Metabolic Dysfunction Associated Fatty Liver Disease
Brief Title: Intermittent Fasting and Metabolic Dysfunction Associated Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Principal Investigator, Tugce Ozlu Karahan, Assistant Professor, Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAFLDIF; 24172 (Other Grant/Funding Number: Health Institutes of Türkiye (TUSEB))
Record Dates: First submitted 2024-10-24; First posted 2024-10-29 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Intermittent Fasting; Metabolic Dysfunction-Associated Fatty Liver Disease
Keywords: Intermittent fasting; fibroblast growth factor 21; autophagy; fatty liver; time-restricted eating
MeSH Terms: conditions — Intermittent Fasting; Fatty Liver

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Energy-restricted diet (Active Comparator): The energy-restricted diet group followed an 8-week long dietary treatment involving 22-25 kcal/kg/day based on ideal body weight.
  Interventions: Other: Energy-restricted dietary intervention
- Energy + time-restricted diet (Experimental): Patients in the energy + time-restricted diet group followed the same dietary intervention and a 16:8 eating pattern where they were instructed to restrict their energy intake to an 8-h time window and not to consume energy-containing foods or drinks during the remaining 16 h.
  Interventions: Other: Energy + time-restricted dietary intervention

INTERVENTIONS:
Other: Energy-restricted dietary intervention — The diets were planned based on current guidelines, manuals, systematic reviews, and meta-analyses published in recent years on MAFLD [5-6, 27-28]. In this diet, carbohydrates constituted 50%-55% of total energy intake, proteins constituted 10%-20%, and fats constituted 25%-35%. The content of the diets was tailored to each patient, considering various factors such as sex, age, and physical activity status.
  Arms: Energy-restricted diet
Other: Energy + time-restricted dietary intervention — Patients in the energy + time-restricted diet group followed the same dietary intervention and a 16:8 eating pattern where they were instructed to restrict their energy intake to an 8-h time window and not to consume energy-containing foods or drinks during the remaining 16 h. Participants were allowed to consume energy-free beverages such as water, coffee, and tea during fasting. The timing of the eating window during the day varied according to participants' lifestyles and habits. However, considering the importance of nocturnal fasting, the eating window in all patients started at 10:00-12:00 in the day and ended at 18:00-20:00 in the evening. The energy-restricted diet group did not follow any time restriction in the planning of main meals and snacks.
  Arms: Energy + time-restricted diet

SUMMARY:
Previous studies have investigated the effect of different dietary patterns on metabolic dysfunction-associated fatty liver disease (MAFLD), for which lifestyle modification remains the primary treatment. The present study sought to determine the effect of intermittent fasting on anthropometric measurements, fibroblast growth factor (FGF)-21, and autophagy markers including autophagy-related protein (ATG)-5 and BECLIN-1 levels, as well as on hepatic steatosis and fibrosis levels in overweight or obese patients with MAFLD to elucidate the efficacy of intermittent fasting in the management of MAFLD. The study included 48 patients diagnosed with MAFLD. Patients were randomly assigned into two groups: 22 received a dietary treatment involving 22-25 kcal/kg/day of energy for 8 weeks (energy-restricted diet group), and 26 followed the same dietary intervention and a 16:8 pattern (energy + time-restricted diet group). The patients were assessed for various parameters at baseline (T0) and at the end of the week 8 (T8). The extent of hepatic steatosis and fibrosis was determined using transient elastography on a FibroScan® device. Serum levels of FGF-21, BECLIN-1, and ATG-5 were determined using enzyme-linked immunosorbent assay.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MAFLD
* Aged 18-65 years
* BMI ≥ 25 kg/m²
* A stable body weight (<5 kg weight loss or gain) over the last 3 months preceding the start of the study
* Signed the informed consent form.

Exclusion Criteria:

* An average daily alcohol consumption >20 g for females and >30 g for males
* Pregnant or lactating women
* Patients with ischemic heart disease or heart failure, chronic inflammatory diseases, chronic viral infections, cancer, moderate-to-severe kidney disease, uncontrolled hypertension, and eating disorders
* Those with a history of bariatric surgery
* Those on insulin due to increased risk of hypoglycemia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 55 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-09-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Gastroenterology, Liver Research Unit, Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Czaja MJ. Function of Autophagy in Nonalcoholic Fatty Liver Disease. Dig Dis Sci. 2016 May;61(5):1304-13. doi: 10.1007/s10620-015-4025-x. Epub 2016 Jan 2. PMID 26725058
- [Result] Itoh N. FGF21 as a Hepatokine, Adipokine, and Myokine in Metabolism and Diseases. Front Endocrinol (Lausanne). 2014 Jul 7;5:107. doi: 10.3389/fendo.2014.00107. eCollection 2014. PMID 25071723
- [Result] Kleinert M, Muller TD. A New FGF21 Analog for the Treatment of Fatty Liver Disease. Diabetes. 2020 Aug;69(8):1605-1607. doi: 10.2337/dbi20-0025. No abstract available. PMID 32690662
- [Result] Byun S, Seok S, Kim YC, Zhang Y, Yau P, Iwamori N, Xu HE, Ma J, Kemper B, Kemper JK. Fasting-induced FGF21 signaling activates hepatic autophagy and lipid degradation via JMJD3 histone demethylase. Nat Commun. 2020 Feb 10;11(1):807. doi: 10.1038/s41467-020-14384-z. PMID 32042044
- [Result] Hydes TJ, Ravi S, Loomba R, E Gray M. Evidence-based clinical advice for nutrition and dietary weight loss strategies for the management of NAFLD and NASH. Clin Mol Hepatol. 2020 Oct;26(4):383-400. doi: 10.3350/cmh.2020.0067. Epub 2020 Jul 17. PMID 32674529
- [Result] Eslam M, Sanyal AJ, George J; International Consensus Panel. MAFLD: A Consensus-Driven Proposed Nomenclature for Metabolic Associated Fatty Liver Disease. Gastroenterology. 2020 May;158(7):1999-2014.e1. doi: 10.1053/j.gastro.2019.11.312. Epub 2020 Feb 8. PMID 32044314

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Energy-restricted Diet | Energy + Time-restricted Diet
Started | 27 | 28
Completed | 22 | 26
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Energy-restricted Diet | Energy + Time-restricted Diet | Total
Number analyzed (Participants) | 22 | 26 | 48
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51.0 [42.7 to 57.2] | 46.0 [40.0 to 55.0] | 49.0 [42.0 to 55.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 10 | 11 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Turkish | 22 | 26 | 48
Region of Enrollment [Number; unit: participants]
  Turkey | 22 | 26 | 48

OUTCOME MEASURES:

1. Primary Outcome: Transient Elastography-Controlled Attenuation Parameter
Description: The extent of hepatic steatosis and fibrosis was determined using transient elastography on a FibroScan® device. All FibroScan measurements were performed following the manufacturer's instructions as specified previously. Hepatic steatosis was defined using controlled attenuation parameter (CAP). The CAP measurement, which indicates steatosis, ranged between 100 and 400 dB/m.
Time Frame: Measurements were taken twice baseline and 8 weeks after the intervention.
Population: The number of participants completing the study in the groups is equal to the analysis population in the data table.
Measure: Median (Inter-Quartile Range); unit: db/m
Arm/Group | Energy-restricted Diet | Energy + Time-restricted Diet
Number analyzed (Participants) | 22 | 26
db/m
  Baseline | 319.5 [296.7 to 371.5] | 343.5 [297.0 to 363.2]
  8 weeks after the Intervention (End) | 291.5 [254.5 to 324.2] | 285.0 [268.2 to 353.7]

2. Primary Outcome: Transient Elastography-Liver Stiffness Measurement
Description: The extent of hepatic steatosis and fibrosis was determined using transient elastography on a FibroScan® device. All FibroScan measurements were performed following the manufacturer's instructions as specified previously. The extent of hepatic steatosis and fibrosis was determined using transient elastography on a FibroScan® device. All FibroScan measurements were performed following the manufacturer's instructions as specified previously. Hepatic fibrosis were defined using liver stiffness measurement (LSM). LSM measurement ranged between 2.5 and 75 kPa.
Time Frame: Measurements were taken twice baseline and 8 weeks after the intervention.
Population: The number of participants completing the study in the groups is equal to the analysis population in the data table.
Measure: Median (Inter-Quartile Range); unit: kpa
Arm/Group | Energy-restricted Diet | Energy + Time-restricted Diet
Number analyzed (Participants) | 22 | 26
kpa
  Baseline | 5.5 [4.2 to 6.2] | 5.7 [4.6 to 6.9]
  8 weeks after the Intervention (End) | 5.1 [4.3 to 6.3] | 4.8 [3.9 to 6.5]

3. Secondary Outcome: Serum Fibroblast Growth Factor-21
Description: At each time point (baseline and week 8), one serum sample was collected per participant. Serum Fibroblast Growth Factor-21 (FGF-21) levels were analyzed using enzyme-linked immunosorbent assay (ELISA) kits, following the manufacturer's protocols (Human FGF-21 ELISA, Biovendor, Czech Republic).
Time Frame: Measurements were taken baseline before and 8 weeks after the intervention.
Population: The number of participants completing the study in the groups is equal to the analysis population in the data table.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Energy-restricted Diet | Energy + Time-restricted Diet
Number analyzed (Participants) | 22 | 26
pg/mL
  Baseline | 316.9 [135.0 to 431.7] | 371.4 [277.7 to 505.1]
  8 weeks after the Intervention (End) | 278.1 [94.8 to 331.6] | 199.1 [109.8 to 459.6]

4. Secondary Outcome: Serum Autophagy-Related Protein-5
Description: At each time point (baseline and week 8), one serum sample was collected per participant. Serum autophagy-related protein-5 (ATG-5) were analyzed using enzyme-linked immunosorbent assay (ELISA) kits, following the manufacturer's protocols (Human Autophagy protein 5 [ATG5] ELISA Kit, MyBioSource, Inc. USA).
Time Frame: Measurements were taken twice baseline and 8 weeks after the intervention.
Population: The number of participants completing the study in the groups is equal to the analysis population in the data table.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Energy-restricted Diet | Energy + Time-restricted Diet
Number analyzed (Participants) | 22 | 26
ng/ml
  Baseline | 0.67 [0.56 to 0.79] | 0.74 [0.46 to 1.29]
  8 weeks after the Intervention (End) | 0.82 [0.48 to 1.01] | 0.95 [0.73 to 1.32]

5. Secondary Outcome: Serum Beclin-1
Description: At each time point (baseline and week 8), one serum sample was collected per participant. Serum Beclin-1 were analyzed using enzyme-linked immunosorbent assay (ELISA) kits, following the manufacturer's protocols (Human BECN1 [Beclin 1] ELISA Kit, ElabScience, USA).
Time Frame: Measurements were taken twice baseline and 8 weeks after the intervention.
Population: The number of participants completing the study in the groups is equal to the analysis population in the data table.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Energy-restricted Diet | Energy + Time-restricted Diet
Number analyzed (Participants) | 22 | 26
ng/ml
  Baseline | 0.18 [0.15 to 0.23] | 0.18 [0.16 to 0.21]
  8 weeks after the Intervention (End) | 0.19 [0.16 to 0.24] | 0.19 [0.15 to 0.20]

ADVERSE EVENTS:
Time Frame: From baseline until end of follow-up, up to 8 weeks
Arm/Group | Energy-restricted Diet | Energy + Time-restricted Diet
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/26
Other Adverse Events (participants affected / at risk) | 0/22 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT06664684/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT06664684/SAP_001.pdf
  • Informed Consent Form (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT06664684/ICF_002.pdf